CLINICAL TRIAL: NCT00291018
Title: A Multi-Center, Prospective, Randomized, Controlled Clinical Trial Comparing the Safety and Effectiveness of ProDisc-C to Anterior Cervical Discectomy and Fusion (ACDF) Surgery in the Treatment of Symptomatic Cervical Disc Disease (SCDD)
Brief Title: Safety and Efficacy Study Comparing ProDisc-C to ACDF Surgery to Treat SCDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDC-08122003
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Symptomatic Cervical Disc Disease
Keywords: ProDisc; ProDisc-C; Spinal Fusion; Anterior cervical diskectomy; Cervical spine; Disc disease; Implant; Degenerative disc disease; Intervertebral disc
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Total Disc Replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ProDisc-C (Experimental): ProDisc-C total disc replacement device intended to treat single level SCDD in the cervical spine from C3-C7
  Interventions: Device: Total Disc Replacement
- Control (Active Comparator): ACDF
  Interventions: Device: ACDF

INTERVENTIONS:
Device: Total Disc Replacement — Total Disc Replacement using ProDisc-C
  Other Names: ProDisc-C
  Arms: ProDisc-C
Device: ACDF — Anterior Cervical Discectomy and Fusion
  Other Names: Control
  Arms: Control

SUMMARY:
The objective of this clinical investigation is to compare the safety and effectiveness of ProDisc-C to anterior cervical discectomy and fusion (ACDF) surgery in the treatment of symptomatic cervical disc disease (SCDD).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cervical disc disease (SCDD) in one vertebral level between C3-C7 defined as: Neck or arm (radicular) pain; and/or a functional/neurological deficit with at least one of the following conditions confirmed by imaging (CT, MRI or X-rays): Herniated nucleus pulposus; Spondylosis (defined by the presence of osteophytes); and/or Loss of disc height.
* Age between 18 and 60 years.
* Unresponsive to non-operative treatment for approximately six weeks or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of conservative treatment.
* NDI score greater than or equal to 15/50 (30%).
* Psychosocially, mentally and physically able to fully comply with the protocol including adhering to follow-up schedule and requirements and filling out forms.
* Signed informed consent.

Exclusion Criteria:

* More than one vertebral level requiring treatment.
* Marked cervical instability on resting lateral or flexion/extension radiographs: translation greater than 3mm and/or greater than 11 degrees of rotational difference to that of either adjacent level.
* Has a fused level adjacent to the level to be treated.
* Radiographic confirmation of severe facet joint disease or degeneration.
* Known allergy to cobalt, chromium, molybdenum, titanium or polyethylene.
* Clinically comprised vertebral bodies at the affected level(s) due to current or past trauma, e.g. by the radiographic appearance of fracture callus, malunion or nonunion.
* Prior surgery at the level to be treated.
* Severe spondylosis at the level to be treated as characterized by any of the following: Bridging osteophytes; A loss of disc height greater than 50%; or Absence of motion (<2°).
* Neck or arm pain of unknown etiology.
* Osteoporosis: A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients who require a DEXA (dual energy x-ray absoptiometry) bone mineral density measurement. If DEXA is required, exclusion will be defined as a DEXA bone density measured T score less than or equal to -2.5 (the World Health Organization definition of osteoporosis).
* Paget's disease, osteomalacia or any other metabolic bone disease (excluding osteoporosis which is addressed above).
* Severe diabetes mellitus requiring daily insulin management.
* Pregnant or interested in becoming pregnant in the next three years.
* Active infection - systemic or local.
* Taking medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids).
* Rheumatoid arthritis or other autoimmune disease.
* Systemic disease including AIDS, HIV, hepatitis.
* Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 368 (Actual)
Dates: Start 2003-08-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

REFERENCES:
- [Derived] Mancuso CA, Cammisa FP, Sama AA, Hughes AP, Girardi FP. Development of an expectations survey for patients undergoing cervical spine surgery. Spine (Phila Pa 1976). 2013 Apr 20;38(9):718-25. doi: 10.1097/BRS.0b013e31827bf204. PMID 23138404
- [Derived] Zigler JE, Delamarter R, Murrey D, Spivak J, Janssen M. ProDisc-C and anterior cervical discectomy and fusion as surgical treatment for single-level cervical symptomatic degenerative disc disease: five-year results of a Food and Drug Administration study. Spine (Phila Pa 1976). 2013 Feb 1;38(3):203-9. doi: 10.1097/BRS.0b013e318278eb38. PMID 23080427

RESULTS

PARTICIPANT FLOW:
Groups:
- ProDisc-C: ProDisc-C total disc replacement device intended to treat single level SCDD in the cervical spine from C3-C7 Total Disc Replacement Randomized Group
- Control: Anterior Cervical Discectomy and Fusion ACDF Randomized Group
- ProDisc-C Continued Access: ProDisc-C total disc replacement device intended to treat single level SCDD in the cervical spine from C3-C7 Total Disc Replacement Non-Randomized Group
Period: Overall Study
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Started | 103 (Enrolled and Treated. 111 PDC subjects were Enrolled but only 103 were Treated.) | 106 (Enrolled and Treated. 117 ACDF subjects were Enrolled but only 106 were Treated.) | 136 (Enrolled and Treated. 140 PDC-CA subjects were Enrolled but only 136 were Treated.)
Evaluated at 24 Months | 99 | 92 | 105
Completed | 78 (Evaluated at 84 Months) | 64 (Evaluated at 84 Months) | 93 (Evaluated at 84 Months)
Not Completed | 25 | 42 | 43
Not completed — Not Consented or Declined PAS | 12 | 15 | 15
Not completed — Death | 3 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 8 | 1
Not completed — Failures | 5 | 12 | 5
Not completed — Lost to Follow-up | 3 | 4 | 18

BASELINE CHARACTERISTICS:
Population: Number of subjects enrolled and treated
Groups:
- ProDisc-C: ProDisc-C total disc replacement device intended to treat single level SCDD in the cervical spine from C3-C7 Total Disc Replacement Randomized
- Control: Anterior Cervical Discectomy and Fusion ACDF Randomized
- ProDisc-C Continued Access: ProDisc-C total disc replacement device intended to treat single level SCDD in the cervical spine from C3-C7 Total Disc Replacement Non-Randomized
- Total: Total of all reporting groups
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access | Total
Number analyzed (Participants) | 103 | 106 | 136 | 345
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (8.42) | 43.5 (7.15) | 43.4 (7.95) | 43.1 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants] — number of subjects who are female or male
  Participants
    Female | 57 | 57 | 78 | 192
    Male | 46 | 49 | 58 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 5
  White | 88 | 97 | 125 | 310
  More than one race | 3 | 5 | 2 | 10
  Unknown or Not Reported | 3 | 3 | 4 | 10
Region of Enrollment [Number; unit: Participants]
  United States | 103 | 106 | 136 | 345
Smoking Status [Number; unit: Subjects]
  Never | 51 | 49 | 79 | 179
  Former | 18 | 20 | 30 | 68
  Current | 34 | 37 | 27 | 98
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (5.32) | 27.3 (5.54) | 26.6 (5.07) | 26.8 (5.29)
Duration of Neck/Arm Pain [Number; unit: Subjects]
  < 6 weeks | 3 | 3 | 1 | 7
  6 weeks to 1 year | 44 | 44 | 49 | 137
  > 1 year | 56 | 59 | 86 | 201

OUTCOME MEASURES:

1. Primary Outcome: Overall Success
Description: Sponsor Definition of Overall Success: (1) Subject's NDI score improved by at least 20% over preoperative baseline value (2) Subject's neurologic parameters, i.e. motor, sensory, and reflexes were maintained or improved as compared to preoperative baseline value (3) No removals, revisions, re-operations, or additional fixation were required to modify any implant (4) No adverse events occurred which were related to the treatment, ProDisc-C or its implantation or ACDF surgery or its associated implants or graft material
Time Frame: 84 Months
Population: Subjects with data at 84 months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 86 | 79 | 102
% of Subjects | 62.8 | 53.2 | 62.7

2. Secondary Outcome: Neurologic Success
Description: % of subjects who were a neurological success (i.e. the patient's neurologic parameters, i.e. motor, sensory, and reflexes are maintained or improved as compared to preoperative baseline value)
Time Frame: 84 months
Population: Subjects who were "per protocol" excluding device failures
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 77 | 64 | 93
% of Subjects | 87.0 | 89.1 | 93.5

3. Secondary Outcome: NDI
Description: NDI is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation and is the most commonly used self-report measure for neck pain.
  The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0-5 rating scale (0='No pain' and 5='Worst imaginable pain'). The points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage: 0 points or 0% means no activity limitations, 50 points or 100% means complete activity limitation.
  Mean duration of the test is 3-8 minutes and the results can be interpreted as:
  * 0-4 points (0-8%) no disability;
  * 5-14 points (10-28%) mild disability;
  * 15-24 points (30-48%) moderate disability;
  * 25-34 points (50-64%) severe disability;
  * 35-50 points (70-100%) complete disability
Time Frame: 84 months
Population: Completed the NDI Questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 64 | 93
% of Subjects
  Significant Improvement (greater than 20% change) | 84.6 | 84.4 | 81.7
  Improvement (3% to 20% change) | 9.0 | 9.4 | 9.7
  No Change (-3% to 3% change) | 1.3 | 0.0 | 3.2
  Deterioration (less than -3% change) | 5.1 | 6.3 | 5.4

4. Secondary Outcome: SF-36 Physical Composite Score (PCS)
Description: The Short form-36 (SF-36) is a 36 item questionnaire which measures Quality of Life (QoL) across eight domains, which are both physically and emotionally based. The eight domains that the SF-36 measures are as follows: physical functioning; role limitations due to physical health; role limitations due to emotional problems; energy/fatigue; emotional well-being; social functioning; pain; general health. A single item is also included that identifies perceived change in health, making the SF-36 a useful indicator for change in QoL over time and treatment.
  It can take patients at least half an hour to complete the SF-36.
  The Physical Composite Score (PCS) specifically looks at the mean average of all of the physically relevant questions.
Time Frame: 84 Months
Population: Subjects who completed the SF-36 questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 62 | 90
% of Subjects
  Significant Improvement (>15% change) | 78.2 | 74.2 | 68.9
  Improvement (3% to 15% change) | 7.7 | 16.1 | 11.1
  No Change (-3% to 3% change) | 2.6 | 3.2 | 2.2
  Deterioration (less than -3% change) | 11.5 | 6.5 | 17.8

5. Secondary Outcome: SF-36 Mental Composite Score (MCS)
Description: The Short form-36 (SF-36) is a 36 item questionnaire which measures Quality of Life (QoL) across eight domains, which are both physically and emotionally based. The eight domains that the SF-36 measures are as follows: physical functioning; role limitations due to physical health; role limitations due to emotional problems; energy/fatigue; emotional well-being; social functioning; pain; general health. A single item is also included that identifies perceived change in health, making the SF-36 a useful indicator for change in QoL over time and treatment.
  It can take patients at least half an hour to complete the SF-36.
  The Mental Composite Score (MCS) specifically looks at the mean average of all of the mental or emotional relevant questions.
Time Frame: 84 Months
Population: Subjects who completed the SF-36 questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 62 | 90
% of Subjects
  Significant Improvement (>15% change) | 52.6 | 50.0 | 54.4
  Improvement (3% to 15% change) | 19.2 | 22.6 | 21.1
  No Change (-3% to 3% change) | 9.0 | 3.2 | 5.6
  Deterioration (less than -3% change) | 19.2 | 24.2 | 18.9

6. Secondary Outcome: VAS Satisfaction
Description: The Visual Analog Scale (VAS) is a commonly used questionnaire and is presented as a 100mm horizontal line. A patient represents their personal opinion regarding their health by adding a vertical line on the VAS horizontal line between the extremes of "No Satisfaction [with the surgery/outcome]" at 0mm and "Complete Satisfaction [with the surgery/outcome]" at 100mm.
Time Frame: 84 Months
Population: Subjects who completed the VAS Satisfaction Questionnaire at 84 Months
Measure: Mean (Standard Deviation)
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 64 | 93
Value | 86.16 (23.750) | 82.09 (29.331) | 86.51 (23.531)

7. Secondary Outcome: VAS Neck Pain Intensity
Description: The Visual Analog Scale (VAS) is a commonly used questionnaire and is presented as a 100mm horizontal line. A patient represents their personal opinion regarding their health by adding a vertical line on the VAS horizontal line between the extremes of "No [Neck] Pain" at 0mm and "Worst [Neck] Pain Possible" at 100mm.
Time Frame: 84 Months
Population: Subjects who completed the VAS Neck Pain Intensity Questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 62 | 93
% of Subjects
  Significant Improvement (more than -20mm change) | 76.9 | 72.6 | 78.5
  Improvement (-3mm to -20mm change) | 10.3 | 14.5 | 17.2
  No Change (-3mm to 3mm change) | 5.1 | 4.8 | 2.2
  Deterioration (more than 3mm) | 7.7 | 8.1 | 2.2

8. Secondary Outcome: VAS Neck Pain Frequency
Description: The Visual Analog Scale (VAS) is a commonly used questionnaire and is presented as a 100mm horizontal line. A patient represents their personal opinion regarding their health by adding a vertical line on the VAS horizontal line between the extremes of "None of the Time [Neck] Pain" at 0mm and "All of the Time [Neck] Pain" at 100mm.
Time Frame: 84 Months
Population: Subjects who completed the VAS Neck Pain Frequency Questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 62 | 93
% of Subjects
  Significant Improvement (more than -20mm change) | 78.2 | 74.2 | 73.1
  Improvement (-3mm to -20mm change) | 10.3 | 11.3 | 12.9
  No Change (-3mm to 3mm change) | 9.0 | 3.2 | 3.2
  Deterioration (more than 3mm) | 2.6 | 11.3 | 10.8

9. Secondary Outcome: VAS Arm Pain Intensity
Description: The Visual Analog Scale (VAS) is a commonly used questionnaire and is presented as a 100mm horizontal line. A patient represents their personal opinion regarding their health by adding a vertical line on the VAS horizontal line between the extremes of "No [Arm] Pain" at 0mm and "Worst [Arm] Pain Possible" at 100mm.
Time Frame: 84 Months
Population: Subjects who completed the VAS Arm Pain Intensity Questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 62 | 93
% of Subjects
  Significant Improvement (more than -20mm change) | 66.7 | 74.2 | 68.8
  Improvement (-3mm to -20mm change) | 16.7 | 9.7 | 15.1
  No Change (-3mm to 3mm change) | 7.7 | 4.8 | 6.5
  Deterioration (more than 3mm) | 9.0 | 11.3 | 9.7

10. Secondary Outcome: VAS Arm Pain Frequency
Description: The Visual Analog Scale (VAS) is a commonly used questionnaire and is presented as a 100mm horizontal line. A patient represents their personal opinion regarding their health by adding a vertical line on the VAS horizontal line between the extremes of "None of the Time [Arm] Pain" at 0mm and "All of the Time [Arm] Pain" at 100mm.
Time Frame: 84 Months
Population: Subjects who completed the VAS Arm Pain Frequency Questionnaire at 84 Months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 61 | 93
% of Subjects
  Significant Improvement (more than -20mm change) | 61.5 | 75.4 | 66.7
  Improvement (-3mm to -20mm change) | 21.8 | 8.2 | 15.1
  No Change (-3mm to 3mm change) | 10.3 | 8.2 | 7.5
  Deterioration (more than 3mm) | 6.4 | 8.2 | 10.8

11. Secondary Outcome: Surgery Again
Description: % of subjects who would opt to have the surgery again if given the choice at 84 months
Time Frame: 84 Months
Population: Subjects who completed this questionnaire at 84 months
Measure: Number; unit: % of Subjects
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Number analyzed (Participants) | 78 | 64 | 92
% of Subjects
  Yes | 92.3 | 81.3 | 91.3
  Maybe | 6.4 | 14.1 | 7.6
  No | 1.3 | 4.7 | 1.1

ADVERSE EVENTS:
Time Frame: 84 Months (i.e. 7 years)
Description: All adverse events were captured from time of consent through the end of study (i.e. 84 Months)
Arm/Group | ProDisc-C | Control | ProDisc-C Continued Access
Serious Adverse Events (participants affected / at risk) | 45/103 | 53/106 | 58/136
Other Adverse Events (participants affected / at risk) | 98/103 | 100/106 | 121/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProDisc-C (N=103) | Control (N=106) | ProDisc-C Continued Access (N=136)
Pain - Back and Lower Extremities (Nervous system disorders) | 6 (7) | 2 (2) | 4 (6)
Pain - Shoulder (Nervous system disorders) | 5 (8) | 4 (4) | 7 (9)
Surgery - Index Level (Surgical and medical procedures) | 2 (2) | 10 (10) | 1 (1) — Surgery at the original index level of the cervical spine
Surgery - Other (Surgical and medical procedures) | 21 (27) | 27 (37) | 18 (29) — Surgery not at the index (cervical level)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 5 (6) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 1 (1)
Pain - Back (Nervous system disorders) | 4 (4) | 3 (4) | 5 (7)
Pain - Neck and Upper Extremities (Nervous system disorders) | 2 (2) | 5 (9) | 2 (2)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1) | 4 (4)
Death (General disorders) | 3 (3) | 3 (3) | 4 (4)
Pain - Neck (Nervous system disorders) | 1 (1) | 3 (3) | 4 (5)
Pain - Other (Nervous system disorders) | 3 (3) | 1 (1) | 3 (4)
Cardiovascular (Cardiac disorders) | 3 (3) | 3 (3) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProDisc-C (N=103) | Control (N=106) | ProDisc-C Continued Access (N=136)
Pain - Neck (Nervous system disorders) | 35 (43) | 41 (62) | 59 (86)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 34 (45) | 22 (31) | 39 (58)
Headaches (Nervous system disorders) | 27 (30) | 21 (23) | 31 (36)
Pain - Back (Nervous system disorders) | 26 (31) | 22 (28) | 32 (57)
Surgery - Other (Surgical and medical procedures) | 23 (30) | 29 (39) | 24 (41) — Surgery not at the index (cervical) level
Pain - Shoulder (Nervous system disorders) | 20 (27) | 22 (24) | 33 (46)
Pain - Upper Extremities (Nervous system disorders) | 20 (27) | 15 (20) | 34 (43)
Gastrointestinal (Gastrointestinal disorders) | 19 (25) | 19 (24) | 14 (20)
Neurological (Psychiatric disorders) | 19 (26) | 15 (16) | 29 (39)
Other (General disorders) | 19 (24) | 18 (24) | 21 (31)
Numbness Non-Index Level Related (Nervous system disorders) | 18 (21) | 15 (17) | 22 (25)
Pain - Back and Lower Extremities (Nervous system disorders) | 18 (33) | 9 (12) | 14 (17)
Pain - Other (Nervous system disorders) | 15 (26) | 17 (19) | 20 (23)
Dysphagia (Nervous system disorders) | 11 (11) | 13 (13) | 15 (19)
Pain - Neck and Upper Extremities with Numbness (Nervous system disorders) | 10 (10) | 10 (17) | 6 (7)
Cardiovascular (Cardiac disorders) | 9 (11) | 11 (12) | 12 (13)
Genitourinary (Renal and urinary disorders) | 8 (8) | 5 (6) | 11 (11)
Insomnia (General disorders) | 8 (8) | 3 (3) | 3 (3)
Pain - Neck and Shoulder (Nervous system disorders) | 8 (9) | 10 (10) | 8 (8)
Pain - Neck and Upper Extremities (Nervous system disorders) | 7 (7) | 22 (30) | 20 (25)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6) | 6 (7)
Infection - Other Non-Wound Related (Infections and infestations) | 6 (7) | 11 (11) | 6 (6)
Pain - Upper Extremities with Numbness (Nervous system disorders) | 6 (7) | 11 (11) | 11 (17)
Musculoskeletal Spasms - Neck (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 12 (12)
Psychological (Psychiatric disorders) | 5 (5) | 11 (12) | 9 (11)
Surgery - Index Level (Surgical and medical procedures) | 2 (2) | 10 (10) | 1 (1) — Surgery at the index level (cervical)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less